CLINICAL TRIAL: NCT03359239
Title: Pilot Study of Atezolizumab Plus PGV001, a Multipeptide Personalized Neoantigen Vaccine, in Patients With Locally Advanced or Metad or Metastatic Urothelial Cancer
Brief Title: Atezolizumab Given in Combination With a Personalized Vaccine in Patients With Urothelial Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Matthew Galsky (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Matthew Galsky, Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 16-1387
Record Dates: First submitted 2017-11-27; First posted 2017-12-02 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Urothelial/Bladder Cancer, Nos
Keywords: PGV001; atezolizumab; urothelial cancer; personalized neoantigen vaccine
MeSH Terms: conditions — Urologic Neoplasms | interventions — atezolizumab; poly ICLC; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PGV 001 with Atezolizumab (Experimental): Atezolizumab: programmed death-ligand 1 PGV001:personalized cancer vaccine PGV 001 - vaccine Poly ICLC- adjuvant The product is prepared within the Icahn School of Medicine at Mount Sinai (ISMMS) . The product consists of two independent preparations of patient specific long peptides mixed with poly-ICLC.
  Interventions: Drug: Atezolizumab; Biological: PGV001; Drug: Poly ICLC; Drug: Normal saline

INTERVENTIONS:
Drug: Atezolizumab — 1200 mg administered by IV infusion every 3 weeks (21 [+/-2] days) for up to 12 months in the adjuvant setting and up to 24 months in the metastatic setting.
  Other Names: TECENTRIQ
Biological: PGV001 — PGV001: up to ten total doses of PGV001with helper peptides. The product is prepared within the ISMMS . The product consists of two independent preparations of patient specific long peptides mixed with poly-ICLC.
  A dose of PGV001 consists of the following:
  Up to ten synthetic peptides - 100μg (0.01 mL, 10 mg/mL) per peptide. One tetanus helper peptide - 100μg (0.01 mL, 10 mg/mL)
Drug: Poly ICLC — 1.4 mg (0.7 mL, 2 mg/mL)
Drug: Normal saline — 0.19 mL

SUMMARY:
The purpose of this study is to determine the good and bad effects of atezolizumab given in combination with a personalized cancer vaccine in patients with urothelial cancer either after surgery to remove organ where the tumor arose (for example, removal of the bladder) or for urothelial cancer that has spread to other organs.

DETAILED DESCRIPTION:
This is a single arm, proof-of-concept study. Fifteen subjects with urothelial cancer interested in participation will sign a "tissue acquisition and vaccine preparation consent" after which tumor tissue will be obtained from either a surgical resection specimen or biopsy. Subjects are scheduled to undergo cystectomy or nephroureterectomy for invasive urothelial cancer may consent prior to, or within 6 weeks after, surgery. The tumor specimen will be submitted for genomic sequencing followed by neoantigen identification utilizing a computational pipeline. Peptides corresponding to these neoantigens will be prepared for the personalized vaccine product. Subjects eligible for the treatment phase of the protocol (i.e., after surgery in adjuvant patients and chemotherapy in metastatic patients) will receive atezolizumab every 3 weeks plus up to ten doses of PGV001 vaccination plus Poly-ICLC. The primary objectives will be to determine the feasibility and safety of administration of a personalized neoantigen-based vaccine (PGV001) plus atezolizumab in subjects with locally advanced or metastatic urothelial cancer.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and HIPAA authorization for release of personal health information.
* Age ≥ 18 years at the time of consent.
* ECOG Performance Status of ≤ 1 within fourteen days of registration for protocol therapy.
* Histological or cytological evidence of urothelial cancer of the bladder, urethra, ureter, or renal pelvis. Differentiation with variant histologies (e.g., squamous cell differentiated) or pure variant histologies will be permitted provided that the predominant histology is urothelial carcinoma.
* Clinical disease state specific criteria:

  * Subjects with invasive urothelial cancer of the bladder or upper urinary tract may consent either before or within 6 weeks after radical cystectomy or nephroureterectomy.
  * Subjects with metastatic and/or unresectable disease must have a metastatic site amenable to biopsy. In situations where a metastatic biopsy does not yield sufficient genetic material for sequencing, or a biopsy cannot be feasibly performed, the use of archival tumor tissue may be considered on a case by case basis. The archival tissue must be derived from a muscle-invasive urothelial cancer specimen or metastatic urothelial cancer specimen.
* Required laboratory values must be obtained within thirty days of consent.

  * ANC ≥ 1500 cells/µL
  * WBC counts > 2500/µL
  * Lymphocyte count ≥ 300/µL
  * Platelet count ≥ 100,000/µL
  * Hemoglobin ≥ 8.0 g/dL
  * Total bilirubin ≤ 1.5 x upper limit of normal (ULN) with the following exception:

    o Patients with known Gilbert disease who have serum bilirubin level ≤ 3 x ULN may be enrolled.
  * AST and ALT ≤ 3.0 x ULN with the following exception:

    o Patients with liver involvement: AST and/or ALT ≤ 5 x ULN
  * Alkaline phosphatase ≤ 2.5 x ULN with the following exception:

    o Patients with documented liver involvement or bone metastases: alkaline phosphatase ≤ 5 x ULN
  * Serum creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 30 mL/min on the basis of the Cockcroft-Gault glomerular filtration rate estimation:
  * (140 - age) x (weight in kg) x (0.85 if female) / 72 x (serum creatinine in mg/dL)
  * INR and aPTT ≤ 1.5 x ULN o This applies only to patients who do not receive therapeutic anticoagulation; patients receiving therapeutic anticoagulation (such as low-molecular-weight heparin or warfarin) should be on a stable dose.

Exclusion Criteria:

* Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis; cirrhosis; fatty liver; and inherited liver disease
* Symptomatic CNS metastases and/or metastases to brain stem, midbrain, pons, medulla, cerebellum, or within 10 mm of the optic apparatus (optic nerves and chiasm) and/or history of intracranial hemorrhage or spinal cord hemorrhage
* Pregnancy, lactation, or breastfeeding
* Known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* History or risk of autoimmune disease, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Bell's palsy, Guillain-Barré syndrome, multiple sclerosis, autoimmune thyroid disease, vasculitis, or glomerulonephritis
* Patients with a history of autoimmune hypothyroidism on a stable dose of thyroid replacement hormone may be eligible.
* Patients with controlled Type 1 diabetes mellitus on a stable insulin regimen may be eligible.
* Patients with eczema, psoriasis, lichen simplex chronicus of vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) are permitted provided that they meet the following conditions:
* History of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest computed tomography (CT) scan

  o History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* History of HIV infection or active hepatitis B (chronic or acute) or hepatitis C infection
* Active tuberculosis
* A known additional primary malignancy that is progressing or requires active treatment. Exceptions include cancers that have undergone potentially curative therapy.
* Medication-Related Exclusion Criteria:

  * Prior treatment with anti-PD-1, or anti-PD-L1 therapeutic antibody or pathway targeting agents
  * No history of severe immune-related adverse effects from anti-CTLA 4 (NCI CTCAE Grade 3 and 4)
  * History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
  * Patients with prior allogeneic bone marrow transplantation or prior solid organ transplantation

Please contact site for other inclusion/exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-05-08 (Actual); Primary Completion 2021-10-12 (Actual); Study Completion 2021-10-12 (Actual)

PRIMARY OUTCOMES:
Number of neoantigens | up to 24 months
  Feasibility parameter: Number of neoantigens identified per subject
Number of peptides synthesized | up to 24 months
  Feasibility parameter: Number of peptides synthesized per subject for vaccination
Vaccine Production time | up to 24 months
  Feasibility parameter:
Proportion of consent to tissue acquisition phase | up to 24 months
  Feasibility parameter: Proportion of subjects who consent to the tissue acquisition phase for whom a vaccine product is prepared
Proportion of subjects eligible for the treatment phase | up to 24 months
  Feasibility parameter: Proportion of subjects eligible for the treatment phase who complete the priming course of vaccination plus atezolizumab
Number of toxicities | up to 24 months
  Safety will be assessed by the frequency of toxicities as assessed by NCI-CTCAE 4.0 criteria

SECONDARY OUTCOMES:
Objective Response Rate | up to 24 hours
  Objective Response Rate by RECIST 1.1 . RECIST: complete response, partial response, stable disease, and progressive disease.
Duration of response | up to 24 months
  The duration of response by RECIST 1.1 and immune-related RECIST criteria in patients with metastatic disease
Time to Progression In Adjuvant patients | up to 24 months
  Time-to-progression in adjuvant patients using RECIST: complete response, partial response, stable disease, and progressive disease
Overall Survival | up to 24 months
  Number of participants living

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Galsky, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Derived] Saxena M, Anker JF, Kodysh J, O'Donnell T, Kaminska AM, Meseck M, Hapanowicz O, Niglio SA, Salazar AM, Shah HR, Kinoshita Y, Brody R, Rubinsteyn A, Sebra RP, Bhardwaj N, Galsky MD. Atezolizumab plus personalized neoantigen vaccination in urothelial cancer: a phase 1 trial. Nat Cancer. 2025 Jun;6(6):988-999. doi: 10.1038/s43018-025-00966-7. Epub 2025 May 9. PMID 40346292